CLINICAL TRIAL: NCT01900041
Title: Multicenter, Randomised, Open Label, Comparative Clinical Study to Evaluate the Superiority, Efficacy and Tolerability of Combination Pantovigar With 2% Minoxidil vs 2% Minoxidil in Women With Female Pattern Hair Loss (Including AGA Ludwig's Type 1-2)
Brief Title: A Study to Evaluate the Superiority, Efficacy and Tolerability of Combination Pantovigar With 2% Minoxidil vs 2% Minoxidil in Women With Female Pattern Hair Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Collaborators: LLC Merz Pharma, Russia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRU20040_4002_1
Record Dates: First submitted 2013-06-27; First posted 2013-07-16 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Female Pattern Hair Loss; Androgenetic Alopecia (AGA); Ludwig Type 1; Ludwig Type 2
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pantovigar + Minoxidil 2% (Experimental): Minoxidil 2% is given as background therapy in both arms
  Interventions: Drug: Pantovigar; Drug: Minoxidil 2% only
- Minoxidil 2% only (Other): Minoxidil 2% is given as background therapy in both arms
  Interventions: Drug: Minoxidil 2% only

INTERVENTIONS:
Drug: Pantovigar — 1 capsule of Pantovigar for oral intake, given three times a day. Duration of treatment: 6 months.
  Arms: Pantovigar + Minoxidil 2%
Drug: Minoxidil 2% only — 1 ML of Minoxidil 2% solution twice a day applied to the scalp. Duration of treatment: 6 months.

SUMMARY:
Pantovigar - a high effective product designed primarily for the treatment of diffuse hair loss in women as well as for the treatment of damaged hair, in the combined therapy can be successfully applied in other types of alopecia.

The purpose of this study is to evaluate efficacy and tolerability of combination therapy Pantovigar plus 2% minoxidil vs 2% minoxidil. To collect tolerability data for combined treatment Pantovigar plus 2% Minoxidil course therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female patient complaint of hair loss and/or hair density reduction for more than 3 months.
* More than 15 % of telogen frontoparietal hair as shown in the phototrichogram.

Exclusion Criteria:

* Symptomatic diffuse alopecia (screening for iron and thyroid function, thyroid stimulating hormon, triiodothyrine, ferritin , total iron-binding capacity)
* Active or history of systemic autoimmune disease, e.g. lupus erythematodes etc.
* Hyperandrogenic alopecia (polycystic ovary syndrome, adrenogenital syndrome, tumors with androgenic activity) (testosterone, prolactin hormone, androstenedione, dehydroepiandrosterone)
* Initiation or termination of hormone therapy within 6 months prior to entering study
* Hormone therapy with androgenic action, e.g. norethisterone etc.
* Pregnancy or lactation within 6 months prior to entering study
* Alopecia areata
* Scarring alopecia
* Treatment with hair promoting agent within 3 months prior to entering study
* Known hair loss after drug intake
* Concomitant use of the drugs causing a hair loss (e.g. aromatase inhibitors, thyreostatics, cytostatics, etc,)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Rate of responders to the treatment | Week 16-20 post baseline
  Assessed by the Investigator using the results photo trichogram (TrichoScience). Responders are defined to fulfill at least one of the following criteria:
  * Reduction in the amount of telogen hair to 15% and below
  * Increasing hair growth density
  * Thickening of average hair diameter
  * Reduction in the amount of vellus hair in comparison with initial indicators

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LLC Merz Pharma, Russia
Locations (2):
- Russia (2):
  - State Scientific Center of Dermatology and Cosmetology, Moscow
  - Moscow Scientific Clinical Center of Dermatology and Cosmetology, Moscow